CLINICAL TRIAL: NCT07252011
Title: Restorative Neurophysiology: Feasibility of "Backup and Restore" Technologies for Brains and Bodies
Brief Title: Restorative Neurophysiology: Backing up and Restoring the Brain (BandR)
Acronym: BandR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Greg Siegle, Professor of Psychiatry, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY25020073
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Adults With Variability in Their Mood
Keywords: mood-variability; brain stimulation; neurofeedback; Positive memory recall; Transcranial alternating current stimulation (tACS); electroencephaolography (EEG)
MeSH Terms: interventions — Transcranial Direct Current Stimulation; Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recall + Stimulation + Neurofeedback (Experimental): Participants will be given their subjective ratings and notes from the first session and asked to recreate how they were feeling at their first session during recall-only blocks. In addition, during neurofeedback and stimulation blocks, they will be given access to technologies for restoring neurophysiological features from the first assessment, including their 1) brain state, 2) facial muscle activity, and 3) heart rate variability. They will be provided with this information and asked to match their previous recordings during the neurofeedback blocks, and stimulated using Transcranial alternating current stimulation (TACS), electromyography (EMG), and vibroacoustic stimulation during the stimulation blocks.
  Interventions: Device: Transcranial alternating current stimulation (tACS); Behavioral: Neuro/biofeedback; Behavioral: Recall; Device: Physiological stimulation

INTERVENTIONS:
Device: Transcranial alternating current stimulation (tACS) — Transcranial alternating current stimulation (tACS) is a widely used non-invasive brain stimulation method. The concept underlying alternating current is to simulate the naturally occurring rhythmic pattern of electrophysiological activity of the brain, which can be detected by electroencephalography (EEG). It involves the application of electrodes onto the scalp, which deliver sinusoidal alternating electric currents.
Behavioral: Neuro/biofeedback — Participants will be shown their their brain EEG recordings and parameters from vocal recordings from their "backup" day, and asked to attempt to use behavioral strategies to match the recording
Behavioral: Recall — Participants will be given their subjective ratings and notes from a journaling interval to use as a target to restore their mood to how they were feeling on the Visit 1 backup day
Device: Physiological stimulation — Facial electrical stimulation, and chest-worn vibroacoustic stimulation will be used to affect facial muscle activity and peripheral physiology to better approximate previously assessed states.

SUMMARY:
Study to examine the extent to which neurophysiological states recorded for a specific person on one day can be induced on a subsequent day

DETAILED DESCRIPTION:
The study will be a single-arm design. It involves a longitudinal design in which subjective, physiological, and brain reactivity will be measured on 3 occasions, between ~2 weeks and ~4 months apart. The first assessment will be on a subjectively "good" day (mood rating above 7/10). The second will be on a subjectively "bad" day (mood rating below 3/10) and the third will be within a week of the second session. At the second and third sessions, participants will work to "restore" their brain state to that of the first assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18-65
* have periods of good and bad moods each lasting at least 2 days

Exclusion Criteria:

* Refusal or inability to provide informed consent
* People who report being in frank psychotic episodes or who say they are unable to stay off psychoactive substances during assessments will be excluded. Because we do not want to return participants to manic states, individuals with bipolar I disorder who report being or appear to be in a manic state at their baseline assessment will also be excluded.
* Inability to complete questionnaires written in English. The justification is that many of the primary analyses involve assessment of change in self-reported symptoms using measures normed in English. Participants must thus be able to read those measures to give valid indications of the extent to which they have responded to the intervention.
* Chronic pain that could be exacerbated by electrical stimulation
* Having difficulties in corrected vision or hearing which would prevent efficient processing of the experimental stimuli
* Having a North American Adult Reading Test (NAART) equivalent full scale IQ < 85
* History of a convulsive disorder
* Presence of any neurologic disorder or medication therapy known to decrease seizure threshold (e.g., brain injury, frequent/severe headaches).
* Participants deemed "not a good fit" for the study for other reasons (such as, but not limited to, continually arriving late or rescheduling, not being a trustworthy historian or accurate reporter of symptoms, being belligerent with study staff, or presenting an active suicide risk) can also be excluded.
* Heart condition
* Current severe Diagnostic and Statistical Manual of Mental Disorders (DSM-V) alcohol or substance use disorder, with the exception of nicotine or caffeine. Clinician will access subjects' alcohol and substance use on a case-by-case to determine whether specific cases of mild or moderate alcohol or substance use would also interfere with the effects of the intervention.
* Those who have metal implants in the vicinity of stimulated areas, or who have electrical implants (e.g., pacemakers, vagus nerve stimulator) will be excluded out of an abundance of caution regarding the safety of electrical stimulation.
* Any metal implant or subcutaneous metal in the face or head

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Mean Change in electroencephalogram (EEG) Activity Across 4 Frequency Bands from Baseline | 4 months
  Change in the cosine of pre- and post- vectors for alpha, beta, theta, and gamma band activity from the first to third session
Mean Change in Happiness Visual Analogue Scale (VAS) Ratings From Baseline | 4 months
  Change in Happiness VAS rating (on a scale from 0-100) from the first to third session

CONTACTS AND LOCATIONS:
Overall Officials: Greg Siegle, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No